CLINICAL TRIAL: NCT02028637
Title: Expression of Toll-Like Receptors 2 and 4 in Asthmatic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Astrid Crespo, Department of Respiratory Medicine, Hospital de la Santa Creu i Sant Pau. Institut d'Investigació Biomédica Sant Pau (IIB Sant Pau). Universitat Autònoma de Barcelona, Department of Medicine. Barcelona Respiratory Network (BRN). Barcelona, Spain., Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 43/2009
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
Keywords: asthma; toll like receptor; innate immunity
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- toll like receptor (TLRs) (Experimental): TLRs are a family of proteins responsible for the recognition of Pathogen-Associated Molecular Patters
  Interventions: Other: TLRs

INTERVENTIONS:
Other: TLRs — Recently it has involved the role of TLR (toll-like receptors) in the pathogenesis of asthma.The possible role that TLRs play in the asthma and its recognition as a new endotype asthma, could open new therapeutic expectations.

SUMMARY:
Introduction: Recently it has involved the role of TLR (toll-like receptors) in the pathogenesis of asthma. TLRs are a family of proteins responsible for the recognition of Pathogen-Associated Molecular Patters (PAMPs). The possible role that TLRs play in IgE-dependent asthma (not eosinophilic) and its recognition as a new endotype asthma, could open new therapeutic expectations.

Objective: To analyze the expression of TLR 2 and 4 in monocytes/ macrophages and neutrophils in peripheral blood and induced sputum from asthmatic patients

DETAILED DESCRIPTION:
The investigators studied patients with asthma. All patients underwent the same day an induced sputum, pulmonary function studies, fractional exhaled nitric oxide, blood total IgE and skin test by prick technique. Asthmatic patients were classified according to the criteria of the GINA 2012. The cellular composition was analyzed by flow cytometry. Expression of TLR2 and TLR4 were analyzed using monoclonal antibodies conjugated with fluorochromes appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Adults with persistent asthma (defined as per the Global INitiative for Asthma Management (GINA) criteria)

Exclusion Criteria:

* If they had a respiratory tract infection or asthma exacerbation within 30 days prior to inclusion
* If they were receiving oral steroids or immunosuppressive treatments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The percentage of neutrophils expressing TLR4 in induced sputum decreases in asthma not eosinophilic | 2 years
  The percentage of neutrophils expressing TLR4 in induced sputum decreases in asthma not eosinophilic (IgEnodep).This could suggest that in this type of asthma the defense mechanism of neutrophils could be altered by decreasing expression of these receptors on their cell surface. This mechanism would still be defined. Probably the respiratory infections play an important role.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Crespo, Principal Investigator — Department of Respiratory Medicine, Hospital de la Santa Creu i Sant Pau. Institut d'Investigació Biomédica Sant Pau (IIB Sant Pau). Universitat Autònoma de Barcelona, Department of Medicine.
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] The ENFUMOSA cross-sectional European multicentre study of the clinical phenotype of chronic severe asthma. European Network for Understanding Mechanisms of Severe Asthma. Eur Respir J. 2003 Sep;22(3):470-7. doi: 10.1183/09031936.03.00261903. PMID 14516137
- [Background] Anderson GP. Endotyping asthma: new insights into key pathogenic mechanisms in a complex, heterogeneous disease. Lancet. 2008 Sep 20;372(9643):1107-19. doi: 10.1016/S0140-6736(08)61452-X. PMID 18805339
- [Background] Weiss ST. Eat dirt--the hygiene hypothesis and allergic diseases. N Engl J Med. 2002 Sep 19;347(12):930-1. doi: 10.1056/NEJMe020092. No abstract available. PMID 12239263
- [Background] Gon Y. Toll-like receptors and airway inflammation. Allergol Int. 2008 Mar;57(1):33-7. doi: 10.2332/allergolint.R-07-157. Epub 2008 Mar 1. PMID 18209505
- [Background] Simpson JL, Grissell TV, Douwes J, Scott RJ, Boyle MJ, Gibson PG. Innate immune activation in neutrophilic asthma and bronchiectasis. Thorax. 2007 Mar;62(3):211-8. doi: 10.1136/thx.2006.061358. Epub 2006 Jul 14. PMID 16844729
- [Background] Crespo-Lessmann A, Juarez-Rubio C, Plaza-Moral V. [Role of toll-like receptors in respiratory diseases]. Arch Bronconeumol. 2010 Mar;46(3):135-42. doi: 10.1016/j.arbres.2009.07.011. Epub 2009 Sep 17. PMID 19765883
- [Background] Vidal S, Bellido-Casado J, Granel C, Crespo A, Plaza V, Juarez C. Flow cytometry analysis of leukocytes in induced sputum from asthmatic patients. Immunobiology. 2012 Jul;217(7):692-7. doi: 10.1016/j.imbio.2011.11.008. Epub 2011 Dec 2. PMID 22204819
- See also: Asthma — http://www.ginasthma.org/.